CLINICAL TRIAL: NCT06807788
Title: Evaluation of Platelet Aggregability in Patients with Takayasu's Arteritis
Acronym: PLATE
Status: Active, not recruiting | Type: Observational
Sponsor: Jose Carlos Nicolau (Other)
Responsible Party: Sponsor-Investigator, Jose Carlos Nicolau, Director of the Acute coronary Unit, University of Sao Paulo
Organization: University of Sao Paulo (Other)
Other Study IDs: SDC: 5859/24/070
Record Dates: First submitted 2025-01-29; First posted 2025-02-04 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Takayasu Arteritis (TAK); Vasculitis, Systemic
Keywords: Platelets; Platelet aggregation; Optical aggregometry
MeSH Terms: conditions — Takayasu Arteritis; Systemic Vasculitis | interventions — Clopidogrel

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Takayasu Arteritis Case Group: 50 patients with Takayasu arteritis
  Interventions: Drug: Clopidogrel
- Healthy Volunteers Control Group: 50 healthy volunteers
  Interventions: Drug: Clopidogrel

INTERVENTIONS:
Drug: Clopidogrel — Clopidogrel 75 mg once a day for 14 days.

SUMMARY:
Inflammatory syndromes in general, and primary vasculitis specifically, present a high risk of cardiovascular involvement. Takayasu arteritis (TAK), for example, presents cardiovascular complications in up to 60% of cases. It is a systemic inflammatory disease that primarily affects large vessels, such as the aorta and its main branches. From a pathophysiological point of view, there are several causes that can lead to an exacerbated increase in cardiovascular risk in this population, including accelerated atherosclerosis, pro-inflammatory action of platelets and significant endothelial dysfunction.

In this context, the present case-control study intends to include 100 individuals (50 with TAK - case group, and 50 healthy volunteers - control group), matched by age and sex in a 1:1 ratio. The main objective of the study is to compare platelet aggregability in patients with TAK against healthy volunteers using the AggRAM® test. Among its secondary objectives is the analysis of platelet aggregability by other methods (Plateletworks, Chronolog, and PPAnalysis).

The study aims to significantly contribute to a better understanding of the potential influence of TAK on platelet aggregation and the response to antiplatelet agents, thereby contributing to a better understanding of the disease, with evident prognostic and therapeutic implications.

ELIGIBILITY:
Inclusion Criteria:

* Patients with TAK, according to the ACR/EULAR 2022 classification criteria (score ≥ 5 out of a total of 20 points) [17]
* Age > 18 years
* Using acetylsalicylic acid
* Agreement to sign the Free and Informed Consent Form (TCLE).

Exclusion Criteria:

* Previous hemorrhagic stroke

  * Use of another antiplatelet agent other than acetylsalicylic acid
  * Active infection or current use of systemic antimicrobial therapy
  * Known platelet dysfunction or platelets <150,000/µL or >450,000/µL
  * Severe illness with life expectancy ≤12 months
  * Known liver disease or coagulation disorder
  * Abuse of illicit drugs or alcohol
  * Dementia, psychiatric condition or any condition that, in the researcher's opinion, prevents participation and follow-up in the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 50 patients with Takayasu arteritis
  50 Healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-10-14 (Actual); Primary Completion 2026-10-14 (Estimated); Study Completion 2027-10-14 (Estimated)

PRIMARY OUTCOMES:
Platelet Aggregation analyzed by optical aggregometry-ADP (AggRAM™- Helena Laboratories) | 14 days
  Compare platelet aggregation analyzed by optical aggregometry-ADP (AggRAM™- Helena Laboratórios) between both groups

SECONDARY OUTCOMES:
Platelet aggregability by AggRAM™ arachidonic acid at baseline; | Baseline
  Avaliation of Platelet aggregability by AggRAM™ arachidonic acid at baseline
Platelet aggregability by AggRAM™ ADP after 14 days of use of Clopidogrel 75 mg/day; | 14 days
  Evaluation of Platelet aggregability by AggRAM™ ADP after 14 days of use of Clopidogrel 75 mg/day;
Platelet aggregability by Plateletworks-ADP at baseline and after 14 days of use of Clopidogrel 75 mg/day | 14 days
  Evaluation of Platelet aggregability by Plateletworks-ADP at baseline and after 14 days of use of Clopidogrel 75 mg/day;
Serum levels of ultrasensitive C-reactive protein (hs-CRP); | Baseline
  Avaliation of Serum levels of ultrasensitive C-reactive protein (hs-CRP)
Serum levels of immature platelets; | Baseline
  Evaluation of Serum levels of immature platelets
Platelet count | Baseline
  Evaluation of Platelet count;
Serum levels of P-Selectin | Baseline
  Evaluation of Serum levels of P-Selectin
Serum levels of interleukin 6 | Baseline
  Evaluation of Serum levels of interleukin 6;
Serum levels of Interleukin 1 | Baseline
  Evaluation of interleukin 1
Serum levels of cholesterol ester transfer proteins; | Baseline
  Evaluation of Serum levels of cholesterol ester transfer proteins;
Serum levels of Lipoprotein(a) (LPa) | Baseline
  Evaluation of Serum levels of Lipoprotein(a) (LPa)

OTHER OUTCOMES:
Subgroup Analysis- Sex | Baseline and 14 days
  Sex (male/female)
Subgroup Analysis- Age | Baseline and 14 days
  Age (≥65 years or < 65 years)
Subgroup Analysis- BDI | Baseline and 14 days
  Body Mass Index (<30 or ≥ 30 kg/m2);
Subgroup Analysis- Diabetes mellitus | Baseline and 14 days
  Diabetes mellitus (presence or not);
Subgroup Analysis- Use of Statins | Baseline and 14 days
  Use of Statins (yes or no)
Subgroup Analysis- Smoking | Baseline and 14 days
  Current smoking (yes or no);
Subgroup Analysis- Use of Nonsteroidal Anti-inflammatory drugs | Baseline and 14 days
  Use of Nonesteroidal ANti-inflammatory drugs ( yes or no)
Subgroup Analysis of Glomerular filtration rate (CKD-EPI) (< 60 mL/min/m2 or ≥ 60mL/min/m2) | Baseline and 14 days
  CKD-EPI (< 60 mL/min/m2 or ≥ 60mL/min/m2)
Subgroup Analysis- Use of immunosuppressive agents | Baseline and 14 days
  Use of immunosuppressive agents ( yes or no)
Subgroup Analysis- Use of Biological agents | Baseline and 14 days
  Use of Biological agents ( yes or no)

CONTACTS AND LOCATIONS:
Locations (1):
- Heart Institute (InCor) / University of São Paulo, São Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Grayson PC, Ponte C, Suppiah R, Robson JC, Gribbons KB, Judge A, Craven A, Khalid S, Hutchings A, Danda D, Luqmani RA, Watts RA, Merkel PA; DCVAS Study Group. 2022 American College of Rheumatology/EULAR Classification Criteria for Takayasu Arteritis. Arthritis Rheumatol. 2022 Dec;74(12):1872-1880. doi: 10.1002/art.42324. Epub 2022 Nov 8. PMID 36349501
- [Background] Alibaz-Oner F, Yurdakul S, Aytekin S, Direskeneli H. Impaired endothelial function in patients with Takayasu's arteritis. Acta Cardiol. 2014 Feb;69(1):45-9. doi: 10.1080/ac.69.1.3011344. PMID 24640521
- [Background] Emmi G, Silvestri E, Squatrito D, Amedei A, Niccolai E, D'Elios MM, Della Bella C, Grassi A, Becatti M, Fiorillo C, Emmi L, Vaglio A, Prisco D. Thrombosis in vasculitis: from pathogenesis to treatment. Thromb J. 2015 Apr 16;13:15. doi: 10.1186/s12959-015-0047-z. eCollection 2015. PMID 25883536
- [Background] Bhandari S, Butt SRR, Ishfaq A, Attaallah MH, Ekhator C, Halappa Nagaraj R, Mulmi A, Kamran M, Karski A, Vargas KI, Lazarevic S, Zaman MU, Lakshmipriya Vetrivendan G, Shahzed SMI, Das A, Yadav V, Bellegarde SB, Ullah A. Pathophysiology, Diagnosis, and Management of Takayasu Arteritis: A Review of Current Advances. Cureus. 2023 Jul 29;15(7):e42667. doi: 10.7759/cureus.42667. eCollection 2023 Jul. PMID 37525862
- [Background] Davi G, Patrono C. Platelet activation and atherothrombosis. N Engl J Med. 2007 Dec 13;357(24):2482-94. doi: 10.1056/NEJMra071014. No abstract available. PMID 18077812
- [Background] Chen Y, Zhong H, Zhao Y, Luo X, Gao W. Role of platelet biomarkers in inflammatory response. Biomark Res. 2020 Aug 2;8:28. doi: 10.1186/s40364-020-00207-2. eCollection 2020. PMID 32774856
- [Background] Sonmez O, Sonmez M. Role of platelets in immune system and inflammation. Porto Biomed J. 2017 Nov-Dec;2(6):311-314. doi: 10.1016/j.pbj.2017.05.005. Epub 2017 Oct 12. PMID 32258788
- [Background] Ucar AK, Ozdede A, Kayadibi Y, Adaletli I, Melikoglu M, Fresko I, Seyahi E. Increased arterial stiffness and accelerated atherosclerosis in Takayasu arteritis. Semin Arthritis Rheum. 2023 Jun;60:152199. doi: 10.1016/j.semarthrit.2023.152199. Epub 2023 Mar 29. PMID 37011578
- [Background] Argyropoulou OD, Protogerou AD, Sfikakis PP. Accelerated atheromatosis and arteriosclerosis in primary systemic vasculitides: current evidence and future perspectives. Curr Opin Rheumatol. 2018 Jan;30(1):36-43. doi: 10.1097/BOR.0000000000000453. PMID 29040156
- [Background] Seyahi E, Ugurlu S, Cumali R, Balci H, Seyahi N, Yurdakul S, Yazici H. Atherosclerosis in Takayasu arteritis. Ann Rheum Dis. 2006 Sep;65(9):1202-7. doi: 10.1136/ard.2005.047498. Epub 2006 Jan 26. PMID 16439439
- [Background] Dos Santos AM, Misse RG, Borges IBP, Gualano B, de Souza AWS, Takayama L, Pereira RMR, Shinjo SK. Increased modifiable cardiovascular risk factors in patients with Takayasu arteritis: a multicenter cross-sectional study. Adv Rheumatol. 2021 Jan 8;61(1):1. doi: 10.1186/s42358-020-00157-1. PMID 33419482
- [Background] Cicco S, Desantis V, Vacca A, Cazzato G, Solimando AG, Cirulli A, Noviello S, Susca C, Prete M, Brosolo G, Catena C, Lamanuzzi A, Saltarella I, Frassanito MA, Cimmino A, Ingravallo G, Resta L, Ria R, Montagnani M. Cardiovascular Risk in Patients With Takayasu Arteritis Directly Correlates With Diastolic Dysfunction and Inflammatory Cell Infiltration in the Vessel Wall: A Clinical, ex vivo and in vitro Analysis. Front Med (Lausanne). 2022 May 16;9:863150. doi: 10.3389/fmed.2022.863150. eCollection 2022. PMID 35652080
- [Background] Dua AB, Kalot MA, Husainat NM, Byram K, Springer JM, James KE, Chang Lin Y, Turgunbaev M, Villa-Forte A, Abril A, Langford C, Maz M, Chung SA, Mustafa RA. Takayasu Arteritis: a Systematic Review and Meta-Analysis of Test Accuracy and Benefits and Harms of Common Treatments. ACR Open Rheumatol. 2021 Feb;3(2):80-90. doi: 10.1002/acr2.11186. Epub 2021 Jan 29. PMID 33512784
- [Background] Keser G, Direskeneli H, Aksu K. Management of Takayasu arteritis: a systematic review. Rheumatology (Oxford). 2014 May;53(5):793-801. doi: 10.1093/rheumatology/ket320. Epub 2013 Oct 4. PMID 24097290
- [Background] Misra DP, Sharma A, Karpouzas GA, Kitas GD. Cardiovascular risk in vasculitis. Best Pract Res Clin Rheumatol. 2023 Mar;37(1):101831. doi: 10.1016/j.berh.2023.101831. Epub 2023 Jun 9. PMID 37302927
- [Background] Mwipatayi BP, Jeffery PC, Beningfield SJ, Matley PJ, Naidoo NG, Kalla AA, Kahn D. Takayasu arteritis: clinical features and management: report of 272 cases. ANZ J Surg. 2005 Mar;75(3):110-7. doi: 10.1111/j.1445-2197.2005.03312.x. PMID 15777385
- [Background] Miloslavsky E, Unizony S. The heart in vasculitis. Rheum Dis Clin North Am. 2014 Feb;40(1):11-26. doi: 10.1016/j.rdc.2013.10.006. PMID 24268007